CLINICAL TRIAL: NCT03987022
Title: "ICE-T" Postoperative Multimodal Pain Regimen Compared to the Standard Regimen in Laparoscopic Gynecologic Surgery: a Randomized Controlled Trial
Brief Title: ICE-T Pain Regimen for Total Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Robert Pollard, MD, Associate Professor of Reproductive Biology, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB18-00920
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Opioid Substitution Treatment
Keywords: Anti-inflammatory agents non-steroidal
MeSH Terms: interventions — Ketorolac; Ketorolac Tromethamine; Analgesics, Opioid; Oxycodone; Acetaminophen; Ibuprofen; Hydromorphone; oxycodone-acetaminophen

STUDY DESIGN:
Intervention Model Description: Enrolled patients were randomized at the end of surgery using sequentially numbered opaque sealed envelopes. A statistician developed the 1:1 mixed block randomization sequence using a random number generator; only the statistician was aware of the sequence. They were randomized to 1 of 2 postoperative pain regimens: ICE-T opioid-sparing regimen or the Standard opioid-centric regimen. The pain regimen protocols began upon PACU discharge. Subjects received their regimens as assigned, except that patients assigned to the ICE-T opioid-sparing group who requested additional narcotic medications prior to postoperative day 4 were prescribed supplemental opioids in addition to their ICE-T regimen medications.
Masking Description: The randomized sequence was masked to all except the statistician who developed the sequence. Upon randomization, the participants, care providers, investigators and outcome assessors were aware of the participant study arm allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- "ICE-T" (Experimental): Regimen #1 "ICE-T" Opioid Sparing Regimen At the end of surgery patients will receive 30mg of intravenous (IV) toradol. Once out of the post anesthesia care unit (PACU) patients will receive
  1. ICE PACKS applied to the surgical sites every hour for 20 minutes Around the clock (ATC) until discharge.
  2. 6 hours from the time of first dose of surgery patients will receive 30mg of IV toradol ATC until discharge.
  3. Once out of the PACU will receive 1 gram of Tylenol per os (PO) every 6 hours for a total of 4 grams daily ATC until discharge
  4. Patients will receive dilaudid 0.2mg IV every 3 hours as needed (PRN) for breakthrough pain.
  5. Patients will be discharged home with (PO) Tylenol and PO toradol as needed (PRN).
  6. If patients requested additional opioids prior to POD4 they were given a supplemental narcotic prescription to ensure adequate pain control
  Interventions: Drug: Ketorolac; Drug: Opioids; Other: Ice Packs; Drug: Tylenol; Drug: Dilaudid Injectable Product
- Standard of Care (Control) (Active Comparator): Regimen #2 STANDARD Postoperative Regimen
  1. Once out of the PACU patients will receive "Standard" postoperative regimen
  2. Motrin 600mg PO every 4 hours PRN pain scale 1-3 pain
  3. Percocet 1 tab PO every 4-6 hours PRN pain scale 4-6 pain
  4. Percocet 2 tabs PO every 7-10 hours PRN pain scale 7-10 pain
  5. Patients will receive dilaudid 0.2mg IV every 3 hours PRN for breakthrough pain.
  6. Patients will be discharged home with Motrin and Percocet for pain PRN.
  Interventions: Drug: Opioids; Drug: Motrin; Drug: Dilaudid Injectable Product; Drug: Percocet 5Mg-325Mg Tablet

INTERVENTIONS:
Drug: Ketorolac — Use of non-steroidal anti-inflammatory drug for pain control postoperatively
  Other Names: Toradol
  Arms: "ICE-T"
Drug: Opioids — Use of narcotic for pain control postoperatively
  Other Names: Oxycodone
Other: Ice Packs — Placement of Ice packs on surgical sites postoperatively
  Arms: "ICE-T"
Drug: Tylenol — Use of pain medication postoperatively
  Other Names: Acetaminophen
  Arms: "ICE-T"
Drug: Motrin — Use of non-steroidal anti-inflammatory drug for pain control postoperatively
  Other Names: Ibuprofen
  Arms: Standard of Care (Control)
Drug: Dilaudid Injectable Product — Use of narcotic for pain control postoperatively
  Other Names: Hydromorphone
Drug: Percocet 5Mg-325Mg Tablet — Use of combination tablet of Tylenol and Oxycodone for pain control postoperatively
  Other Names: Oxycodone-Acetaminophen
  Arms: Standard of Care (Control)

SUMMARY:
The purpose of this randomized controlled trial is to determine whether, "ICE-T," a multimodal postoperative pain regimen composed of around the clock ice packs, toradol, and tylenol, has improved pain control compared to the standard narcotic based postoperative pain regimen in patients undergoing total laparoscopic gyn surgery.

DETAILED DESCRIPTION:
Laparoscopy is a frequently used route for hysterectomy. Yet few studies have investigated opioid-sparing postoperative regimens for this common surgery. The study objective was to determine whether ice packs, Tylenol, and Toradol (ICE-T), an opioid-sparing multimodal postoperative pain regimen, has improved pain control compared with a standard opioid-centric postoperative pain regimen in total laparoscopic hysterectomy patients.

The study was a randomized controlled trial. It included total laparoscopic hysterectomy postoperative patients that were randomized to the ICE-T or standard regimen. The ICE-T regimen prescribed scheduled around-the-clock ice-packs, acetaminophen and ketorolac. The standard protocol prescribed as needed ibuprofen and acetaminophen/oxycodone based on pain score. Both regimens included intravenous hydromorphone for breakthrough pain. However, subjects in the ICE-T group who requested additional narcotic medications prior to postoperative day 4, were prescribed supplemental narcotics in addition to the ICE-T regimen. The subjects pain control and quality of recovery were assessed on postoperative day 1 and 4.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are the following:

* Consenting, English speaking women between ages 18 and 80 who will undergo same day laparoscopic gyn surgery at MetroHealth Medical Center
* Ability to read VAS Scores
* Specific procedures include, but are not limited to:

  * Laparoscopic hysterectomy, for uterus 250 g or less
  * Laparoscopic hysterectomy, for uterus 250 g or less; with removal of tube(s), and/or ovary(s)
  * Laparoscopic hysterectomy, for uterus 250 g or less; with removal of tube(s), and/or ovary(s), with repair of enterocele
  * Laparoscopic hysterectomy, for uterus 250 g or less; with repair of enterocele
  * Laparoscopic hysterectomy, for uterus greater than 250 g
  * Laparoscopic hysterectomy, for uterus greater than 250 g; with removal of tube(s) and/or ovary(s)
  * Laparoscopic hysterectomy, for uterus greater than 250 g; with removal of tube(s) and/or ovary(s), with repair of enterocele
  * Laparoscopic hysterectomy, for uterus greater than 250 g; with repair of enterocele

Exclusion Criteria:

* History of chronic pelvic pain
* Abdominal surgery
* History of psychiatric disease
* Currently taking analgesic medications
* Currently taking sedatives
* Liver disease
* Renal disease with CrCl < 60cc/min.
* History of burns from application of ice.
* Women who did not consent for the study.
* Intraoperative concern for increased blood loss
* Unable to speak English
* Unable to understand VAS Scores
* Undergoing concomitant abdominal procedures.
* Allergy to motrin, toradol, Percocet, Tylenol
* Active or history of peptic ulcer disease
* History of GI bleeding or perforation
* Hemorrhagic diathesis
* Severe uncontrolled heart failure
* Inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pollard, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Multimodal opioid-sparing postoperative pain regimen compared with the standard postoperative pain regimen in vaginal pelvic reconstructive surgery: a multicenter randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/31201808/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to surgery, patients will be asked to participate in the study in their private patient rooms or in medical clinic.
Pre-assignment Details: 111 patients were assessed for eligibility, but 45 were excluded (30 did not meet inclusion criteria, and 15 declined to participate). Therefore, 66 patients were randomized.
Groups:
- "ICE-T" Opioid Sparing Regimen: At the end of surgery patients will receive 30mg of intravenous (IV) toradol. Once out of the post anesthesia care unit (PACU) patients will receive
  1. ICE PACKS applied to the surgical sites every hour for 20 minutes Around the clock (ATC) until discharge.
  2. 6 hours from the time of first dose of surgery patients will receive 30mg of IV toradol ATC until discharge.
  3. Once out of the PACU will receive 1 gram of Tylenol per os (PO) every 6 hours for a total of 4 grams daily ATC until discharge
  4. Patients will receive dilaudid 0.2mg IV every 3 hours as needed (PRN) for breakthrough pain.
  5. Patients will be discharged home with (PO) Tylenol and PO toradol as needed (PRN).
- STANDARD Postoperative Regimen: Once out of the PACU patients will receive "Standard" postoperative regimen, which includes:
  1. Motrin 600mg PO every 4 hours PRN pain scale 1-3 pain
  2. Percocet 1 tab PO every 4-6 hours PRN pain scale 4-6 pain
  3. Percocet 2 tabs PO every 7-10 hours PRN pain scale 7-10 pain
  4. Patients will receive dilaudid 0.2mg IV every 3 hours PRN for breakthrough pain.
  5. Patients will be discharged home with Motrin and Percocet for pain PRN.
Period: Overall Study
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Started | 36 | 30
Completed | 33 | 28
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 66 participants were enrolled at baseline (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
Groups:
- ICE-T: Toradol and Tylenol were given as pain management post-operative of total laparoscopic hysterectomy
- Standard of Care (Control): Received routine pain management postoperative of laparoscopic hysterectomy
- Total: Total of all reporting groups
Arm/Group | ICE-T | Standard of Care (Control) | Total
Number analyzed (Participants) | 36 | 30 | 66
Age, Categorical [Count of Participants; unit: Participants] — Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 36 | 30 | 66
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  Participants
    Female | 36 | 30 | 66
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  Participants
    Hispanic or Latino | 4 | 0 | 4
    Not Hispanic or Latino | 32 | 30 | 62
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 19 | 18 | 37
    White | 11 | 11 | 22
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 4 | 0 | 4
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] — Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  kg/m^2 | 31.0 [25.6 to 36.3] | 29.8 [24.4 to 35.3] | 30.8 [25.0 to 35.5]
Depression/Anxiety [Count of Participants; unit: Participants] — Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  Participants | 1 | 1 | 2
Current Smoker [Count of Participants; unit: Participants] — Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  Participants | 7 | 9 | 16
Charlson Comorbidity Index [Median (Inter-Quartile Range); unit: Index] — The Charleston Comorbidity Index calculates the 10-year survival of a patient. It considers age, history of: myocardial infarction, congestive heart failure, peripheral vascular disease, stroke, dementia, chronic obstructive pulmonary disease, connective tissue disease, peptic ulcer disease, liver disease, diabetes mellitus, hemiplegia, chronic kidney disease, solid cancers, leukemia, lymphoma, and AIDS. As this value ranges from 0-37, with highest value of 37 representing 0% survival in 10 years, and lowest value of 0 at 98% survival in 10 years, it is possible for median/mean to be zero. Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  Index | 0 [0 to 0] | 0 [0 to 1] | 0 [0 to 1]
STOP-BANG Score [Median (Inter-Quartile Range); unit: scores on a scale] — The STOP-BANG Score is questionnaire that screens for obstructive sleep apnea. It is an acronym for Snoring, Tiredness, Observed apnea, Pressure (high blood pressure), Body Mass Index, Age greater than 50 years, Neck circumference greater than 40 cm, Gender male (male gender gives an additional score). The score ranges from 0 - 8, with 8 being the highest risk for moderate to severe apnea. Patients are considered to be considered high risk for sleep apnea when their summed score is greater than or equal to 3. Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
  scores on a scale | 1.0 [0.0 to 2.0] | 1.0 [0.0 to 2.0] | 1.0 [0.0 to 2.0]

OUTCOME MEASURES:

1. Primary Outcome: POD1 Visual Analog Pain (VAS) Score
Description: Visual Analog Scores (VAS) Scores in the morning of post op day 1 (~24 hours after surgery) The scale is from 0 to 10 (0=no pain and 10=being worst pain ever)
Time Frame: Morning of post operative day 1 (~24 hours after surgery)
Population: This population are participants that are approximately 24 hours post Total Laparoscopic Hysterectomy procedure. 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up).
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Groups:
- "ICE-T" Opioid Sparing Regimen: At the end of surgery patients will receive 30mg of intravenous (IV) toradol. Once out of the post anesthesia care unit (PACU) patients will receive
  1. ICE PACKS applied to the surgical sites every hour for 20 minutes Around the clock (ATC) until discharge.
  2. 6 hours from the time of first dose of surgery patients will receive 30mg of IV toradol ATC until discharge.
  3. Once out of the PACU will receive 1 gram of Tylenol per os (PO) every 6 hours for a total of 4 grams daily ATC until discharge
  4. Patients will receive dilaudid 0.2mg IV every 3 hours as needed (PRN) for breakthrough pain.
  5. Patients will be discharged home with (PO) Tylenol and PO toradol as needed (PRN).
  6. If patient's requested additional opioids prior to POD4 they were given a supplemental narcotic prescription to ensure adequate pain control
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Number analyzed (Participants) | 32 | 28
Score on a scale | 5.8 [3 to 7] | 5 [3 to 6]
Statistical Analysis 1: Comparison: STANDARD Postoperative Regimen; Test type: Superiority; p = .16, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: POD1 Quality of Recovery Score
Description: QoR-40 is a quality of recovery 40-item questionnaire based on how the patient has felt in the past 24 hours. It provides a global score and sub scores across five dimensions: patient support, comfort, emotions, physical independence, and pain; each item is graded on a five-point Likert scale. QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery). It is a measure of postoperative quality of recovery in a range of clinical and research situations.
Time Frame: Postoperative Day 1
Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 1 outcomes included 60 subjects (n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up).
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Groups:
- "ICE-T" Opioid Sparing Regimen: At the end of surgery patients will receive 30mg of intravenous (IV) toradol. Once out of the post anesthesia care unit (PACU) patients will receive
  1. ICE PACKS applied to the surgical sites every hour for 20 minutes Around the clock (ATC) until discharge.
  2. 6 hours from the time of first dose of surgery patients will receive 30mg of IV toradol ATC until discharge.
  3. Once out of the PACU will receive 1 gram of Tylenol per os (PO) every 6 hours for a total of 4 grams daily ATC until discharge
  4. Patients will receive dilaudid 0.2mg IV every 3 hours as needed (PRN) for breakthrough pain.
  5. Patients will be discharged home with (PO) Tylenol and PO toradol as needed (PRN).
  6. If patients requested additional opioids prior to POD4 they were given a supplemental narcotic prescription to ensure adequate pain control
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Number analyzed (Participants) | 32 | 28
Score on a scale | 161.5 [147.5 to 179.0] | 162.5 [155.0 to 179.5]
Statistical Analysis 1: Comparison: STANDARD Postoperative Regimen; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: 1st 24hr Total Dose of Narcotic
Description: Total amount of narcotic in morphine equivalents administered to patients who were admitted for overnight extended recovery and/or observation. This includes narcotics given intra-operatively, in the post-anesthesia care unit and during their inpatient stay up until 24 hours postop.
Time Frame: Total narcotic use from intra-op to 24 hours post-op
Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The postoperative day 1 analysis outcomes included n= 32 ICE-T arm POD1 analysis, 1 withdrew, 3 loss to follow up; n=28 Standard care arm POD1 analysis, 2 loss to follow up. The subjects who chose same-day discharge were excluded from the analysis of total narcotic use within 24 hours post-op due to differences in reporting and access to medications. The analysis of this variable included n=27 ICE-T arm and n=23 Standard arm.
Measure: Median (Inter-Quartile Range); unit: oral morphine milligram equivalents
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Number analyzed (Participants) | 27 | 23
oral morphine milligram equivalents | 77 [54.3 to 101.0] | 111.5 [84.8 to 121.3]
Statistical Analysis 1: Comparison: STANDARD Postoperative Regimen; Test type: Superiority; p = .01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Length of Stay
Description: Length of hospital stay measured in the number of nights spent at the hospital. Subjects were given the option for same-day discharge home from the PACU or overnight inpatient observation.
Time Frame: Post-operative Day 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: nights
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Number analyzed (Participants) | 32 | 28
nights | 1 [1 to 1] | 1 [1 to 1]
Statistical Analysis 1: Comparison: STANDARD Postoperative Regimen; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: POD4 VAS Scores
Description: Visual Analog Scores 4 days post-surgery. VAS pain score of 0 to a score of worst pain indicating a score of 10 (0=no pain and 10=being worst pain ever)
Time Frame: VAS Scores at 4 days post-surgery.
Population: 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Number analyzed (Participants) | 29 | 23
Score on a scale | 3 [1.5 to 5] | 4 [2.5 to 5]
Statistical Analysis 1: Comparison: STANDARD Postoperative Regimen; Test type: Superiority; p = .58, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: POD4 Quality of Recovery
Description: as for outcome 2
Time Frame: Postoperative Day 4
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Number analyzed (Participants) | 29 | 23
Score on a scale | 179.5 [164.5 to 190.5] | 177.0 [168.0 to 190.0]
Statistical Analysis 1: Comparison: STANDARD Postoperative Regimen; Test type: Superiority; p = .47, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: POD4 Satisfaction Score
Description: Patient's satisfaction with their pain management as of postoperative day 4, rated on a scale of 1 - 10, where 1 is very dissatisfied and 10 is very satisfied.
Time Frame: Data collected as of postoperative day 4
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Groups:
- ICE-T: At the end of surgery patients will receive 30mg of intravenous (IV) toradol. Once out of the post anesthesia care unit (PACU) patients will receive
  1. ICE PACKS applied to the surgical sites every hour for 20 minutes Around the clock (ATC) until discharge.
  2. 6 hours from the time of first dose of surgery patients will receive 30mg of IV toradol ATC until discharge.
  3. Once out of the PACU will receive 1 gram of Tylenol per os (PO) every 6 hours for a total of 4 grams daily ATC until discharge
  4. Patients will receive dilaudid 0.2mg IV every 3 hours as needed (PRN) for breakthrough pain.
  5. Patients will be discharged home with (PO) Tylenol and PO toradol as needed (PRN).
  6. If patients requested additional opioids prior to POD4 they were given a supplemental narcotic prescription to ensure adequate pain control
- Standard of Care (Control): 1. Once out of the PACU patients will receive "Standard" postoperative regimen
  2. Motrin 600mg PO every 4 hours PRN pain scale 1-3 pain
  3. Percocet 1 tab PO every 4-6 hours PRN pain scale 4-6 pain
  4. Percocet 2 tabs PO every 7-10 hours PRN pain scale 7-10 pain
  5. Patients will receive dilaudid 0.2mg IV every 3 hours PRN for breakthrough pain.
  6. Patients will be discharged home with Motrin and Percocet for pain PRN.
Arm/Group | ICE-T | Standard of Care (Control)
Number analyzed (Participants) | 29 | 23
Score on a scale | 10.0 [5.8 to 10.0] | 8.0 [6.0 to 10.0]
Statistical Analysis 1: Comparison: Standard of Care (Control); Test type: Superiority; p = 0.4, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Time to First Bowel Movement
Description: Time to first bowel movement in days
Time Frame: Up to post op day 4
Population: Patients that have undergone procedure were observed to see when they had their first bowel movement post-operation up to 4 days. 66 participants were enrolled (36 ICE-T arm; 30 Standard Care arm). The final analysis for postoperative day 4 outcomes included 52 subjects (n=29 ICE-T arm POD4 analysis, 1 withdrew, 6 loss to follow up; n=23 Standard arm POD4 analysis, 7 loss to follow up).
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Number analyzed (Participants) | 29 | 23
days | 2 [1 to 3] | 3 [2 to 4]
Statistical Analysis 1: Comparison: STANDARD Postoperative Regimen; Test type: Superiority; p = .02, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Oxycodone 5mg Doses Taken Since Discharge
Description: The number of oxycodone 5mg doses (whether as oxycodone 5mg or as percocet 5/325) taken since discharge up until postoperative 4.
Time Frame: Data collected as of Postoperative day 4
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: Doses
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
Number analyzed (Participants) | 29 | 23
Doses | 0 [0.0 to 1.0] | 7.0 [3.0 to 12.0]
Statistical Analysis 1: Comparison: STANDARD Postoperative Regimen; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

10. Other Pre Specified Outcome: "ICE-T" Arm Patients Who Requested Supplemental Narcotics in Addition to Their ICE-T Regimen
Description: Enrolled patients were randomized at the end of surgery to 1 of 2 postoperative pain regimens: ICE-T opioid-sparing regimen or the Standard opioid-centric regimen. The pain regimen protocols began upon PACU discharge. Subjects received their regimens as assigned, except that patients assigned to the ICE-T opioid-sparing group who requested additional narcotic medications prior to postoperative day 4 were prescribed supplemental opioids in addition to their ICE-T regimen medications.
Time Frame: Up until postoperative day 4
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | "ICE-T" Opioid Sparing Regimen
Number analyzed (Participants) | 29
Participants | 8

ADVERSE EVENTS:
Time Frame: Follow up was until postoperative day 4 (POD 4)
Description: Adverse event data was collected from the time of operation up to postoperative day 4. This was systematically collected via chart review, as well as a questionnaire administered to patients via phone in order to capture any events treated outside the study institution.
Arm/Group | "ICE-T" Opioid Sparing Regimen | STANDARD Postoperative Regimen
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/30
Other Adverse Events (participants affected / at risk) | 7/36 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | "ICE-T" Opioid Sparing Regimen (N=36) | STANDARD Postoperative Regimen (N=30)
Intraoperative Complication: Cystotomy (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) — An injury to the bladder during the surgery. The occurrences of these injuries happened prior to the patients randomization in the study.
Emergency Room Visit Post-Operatively - Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Postoperative constipation requiring an emergency room visit
Emergency Room Visit Post-operatively - Pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Uncontrolled postoperative pain requiring an emergency room visit
Emergency Room Visit - Intraoperative complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) — Emergency room visit for urgent follow up on an intraoperative complication
Intraoperative complication: bowel repair (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — An injury to the bowel during the surgery that required repair. The occurrence of this injury happened prior to the patients randomization in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT03987022/Prot_SAP_002.pdf
  • Informed Consent Form (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT03987022/ICF_001.pdf